CLINICAL TRIAL: NCT03804216
Title: Multimodal Imaging Analysis, SD-OCT and OCT Angiography, Retinal Variations Observed in Dialysis Patients
Acronym: OCTADIAL
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: OCTADIAL
Record Dates: First submitted 2019-01-11; First posted 2019-01-15 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Renal Failure
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Multimodal Imaging Analysis — The patients are seen in consultation ophthalmological before and the 1 hour after their session of dialysis. THE OCT angiography and other not invasive ophthalmological examinations will be realized during the follow-up
  Other Names: SD-OCT and OCT Angiography

SUMMARY:
Little knowledge exist on the short and long-term ophthalmological effect of the dialysis. Some studies stated a variation of the thickness subfoveal choroidal before and after a session of dialyse as well as variations of the coat of optical fibers measured in OCT.

The Optical Coherence Tomography angiography OCT is a not invasive imaging technique which is now a part of examinations of investigation in imaging of retina. This technique allows to study the retinal macula vascularization without injection of contrast agent and thus allows to deepen the knowledge in medical domains where the exploration was to limited because of the invasive character of the examinations.

The hypothesis of this project is that hemodynamic change during the hemodialysis may lead fine variations of the retinal vascularization in the short-term (the day of the dialysis) but also in the longer term (over 1 year).

ELIGIBILITY:
Inclusion Criteria:

* Indication of treatment by hemodialysis
* First session of dialysis
* Hemodialysis planned for 1 minimum year

Exclusion Criteria:

* particular ophthalmological Histories: vitreo-retinal surgery, strong nearsightedness, chronic glaucoma
* Unaffiliated in a national insurance scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients in hemodialysis.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-02-26 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
vascular density before hemodialysis | before hemodialysis
  Analysis of the variation of the vascular densities in retinal macula in the central 6 mm
vascular density 1 hour after hemodialysis | 1 hour after hemodialysis
  Analysis of the variation of the vascular densities in retinal macula in the central 6 mm

SECONDARY OUTCOMES:
vascular density 1 month after dialysis | 1 month after dialysis
  Analysis of the variation of the vascular densities in retinal macula in the central 6 mm
vascular density 3 month after dialysis | 3 month after dialysis
  Analysis of the variation of the vascular densities in retinal macula in the central 6 mm
vascular density 6 month after dialysis | 6 month after dialysis
  Analysis of the variation of the vascular densities in retinal macula in the central 6 mm
vascular density 12 month after dialysis | 12 month after dialysis
  Analysis of the variation of the vascular densities in retinal macula in the central 6 mm
vascular density before dialysis | before dialysis
  mesure by OCTA
vascular density 1 hour after dialysis | 1 hour after dialysis
  mesure by OCTA
vascular density 1 month after dialysis | 1 month after dialysis
  mesure by OCTA
vascular density 3 month after dialysis | 3 month after dialysis
  mesure by OCTA
vascular density 6 month after dialysis | 6 month after dialysis
  mesure by OCTA
vascular density 12 month after dialysis | 12 month after dialysis
  mesure by OCTA
size of coat retinal optical fibers before dialysis | before dialysis
  variation of the coat
size of coat retinal optical fibers 1 hour after dialysis | 1 hour after dialysis
  variation of the coat
size of coat retinal optical fibers 1 month after dialysis | 1 month after dialysis
  variation of the coat
size of coat retinal optical fibers 3 month after dialysis | 3 month after dialysis
  variation of the coat
size of coat retinal optical fibers 6 month after dialysis | 6 month after dialysis
  variation of the coat
size of coat retinal optical fibers 12 month after dialysis | 12 month after dialysis
  variation of the coat

CONTACTS AND LOCATIONS:
Locations (1):
- Ophtalmology department, Créteil, France